CLINICAL TRIAL: NCT03454321
Title: Is the Presence of Subacromial Bursitis Associated With a Good Response to Ultrasound-guided Steroid Injection in Rotator Cuff Tendinopathy?
Brief Title: IS'ECHO : Impact of Bursitis on the Efficacy of Subacromial Steroid Injection in Rotator Cuff Tendinopathy
Acronym: IS'ECHO
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0496
Record Dates: First submitted 2018-02-13; First posted 2018-03-05 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: Rotator cuff tendinopathy; ultrasound; subacromial bursitis; steroid injection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Infiltration — The subacromial injection will be performed under ultrasound guidance to accurately inject the subacromial bursae. After skin disinfection with povidone, the injection will be performed with a 21G needle. The bursae will be injected with 2 ml of lidocaine 2% and 1 ml of betamethasone.

SUMMARY:
Shoulder pain is a common reason for medical consultation affecting 6.7 % of the adults from 50 to 70 years old and until 21 % of the adults over 70. Among these painful shoulders, rotator cuff tendinopathy represents 44 to 65% of these consultations. To treat this condition, patients usually receive analgesics and physical therapy. When these treatments are not effective, a corticosteroid sub-acromial injection is proposed. However, according to the literature, there is only about 50% of good response to this subacromial injection in rotator cuff tendinopathy. It has been suggested that the injection could be more effective in the presence of an inflammation over the tendons called bursitis. However, no studies have clearly established this. The objective of the study is to determine if the presence of a bursitis could be a factor of good response to corticosteroid injection. The results could allow us to determine which patients have the best profile to respond to subacromial injection. The investigators hope that these data would improve the treatment of this frequent disease.

DETAILED DESCRIPTION:
Patients referred to receive a subacromial ultrasound-guided injection for shoulder pain related to a rotator cuff tendinopathy will be enrolled in the study. After validation of the inclusion criteria, the participants will receive oral information about the protocol. Then, they will be examined and will undergo X-rays and an ultrasound of their shoulder. Pain shoulder and shoulder disability will be assessed before the injection with a visual analogic pain scale and the Oxford Shoulder Score questionnaire, respectively.

The subacromial injection will be performed under ultrasound guidance to accurately inject the subacromial bursae. After skin disinfection with povidone, the injection will be performed with a 21G needle. The bursae will be injected with 2 ml of lidocaine 2% and 1 ml of betamethasone.

After the procedure, the participants will all receive a standardized physiotherapy.

For primary outcome, the therapeutic response will be assessed 3 months after the procedure. Patients will be considered as having a good response if their level of pain decreases by over 30%.

The number of participants having a good clinical response will be compared between the patients presenting a bursitis and those without bursitis. The comparison will be made using a Chi-2 test.

Others parameters will be studied: reduction in pain 6 weeks after the injection, reduction in shoulder disability 6 weeks and 3 months after the injection. Other ultrasound lesions will be collected so as X-ray features to search other factors associated with the presence or absence of a good therapeutic response (details in secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Major patients with manifestations of rotator cuff tendinopathy referred to our rheumatology department to receive an ultrasound-guided subacromial injection.

Exclusion Criteria:

* Patients refusing to participate
* Allergic to local anesthetics
* Shoulder involvement of an inflammatory rheumatic disease
* History of shoulder surgery
* Shoulder instability
* Glenohumeral osteoarthritis
* Frozen shoulder
* Extended rotator cuff tear
* Tendinous calcification > 0.5 cm
* Pregnant women
* Minors
* Majors under guardianship
* Patient inappropriate for entry into this study according to the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will receive a subacromial ultrasound-guided injection for shoulder pain related to a rotator cuff tendinopathy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Reduction in shoulder pain 3 months after the subacromial corticosteroid injection | 3 months
  The primary outcome is the presence of a therapeutic response 3 months after the intervention. The level of pain will be assessed by a visual analogic pain scale of 0 (absence of pain) to 10 centimeters (maximal pain).
  Participants will be considered as good responders if their level of pain decreases more than 30 percent.
  Safety issue: No

SECONDARY OUTCOMES:
Reduction in shoulder pain 6 weeks after the subacromial steroid injection. | 6 weeks after the intervention
  Presence of a therapeutic response 6 weeks after the intervention considering the reduction in pain between day 0 and Week 6 and assessed with the same scale as the primary outcome. Participants will be considered as good responders if their level of pain decreases more than 30 percent.
Reduction in OSS score (Oxford Shoulder Score) 6 weeks and 3 months after the injection | data from Day 0, Week 6 and Month 3
  The OSS is a 12-item shoulder-specific questionnaire that was developed, with patients, for the assessment of shoulder pain and function. Items refer to the past 4 weeks and each offers five ordinal response options. These were scored from 1 to 5 (5 = most severe) and then conbined to produce a single score with a range from 12 (least difficulties) to 60 (most difficulties).
Presence of other ultrasound lesions associated with a good response to steroid injection | data from Day 0, Week 6 and Month 3
  The ultrasound lesions collected just before the injection will be :
  * Bursitis: the bursitis is defined by a thickening of more than 2 mm of the subacromial bursae.
  * Tendinous lesions (supra-spinatus, infra-spinatus or sub-scapularis): tendon thickening, hypoechoic density, presence of microcalcification, partial or complete tear
  * Effusion of long head of biceps tendon sheath
  * Acromio-clavicular joint lesions = synovitis, presence of Doppler flow, osteophytes
Presence of radiographic abnormalities associated with a good response. | data from Day 0, Week 6 and Month 3
  X-ray data = Acromion Morphology according to Park's classification, Critical Shoulder Angle, acromioclavicular osteoarthritis
Steroid injection safety | data from Day 0, Week 6 and Month 3
  Adverse events will be collected after the procedure and during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Darrieutort-Laffite, Principal Investigator — Nantes University Hospital
Locations (1):
- Chu de Nantes, Nantes, France